CLINICAL TRIAL: NCT00722644
Title: Cognitive Behavioral Treatment of HIV+ Drug Abusers
Brief Title: Cognitive Behavioral Stress Management for HIV+ Drug Abusers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA13802
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-07

CONDITIONS: HIV/AIDS; Drug Abuse; Alcohol Abuse
Keywords: HIV; Medication Adherence; Stress Management; CD4/Viral Loads; Cognitive Behavioral Treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Alcoholism; Medication Adherence

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management

SUMMARY:
The primary purpose of this 5-year study is to determine whether a Cognitive Behavioral Stress Management (CBSM) intervention, demonstrated to be effective in reducing distress, enhancing coping, and maintaining health among HIV+ non-drug abusers (see Schneiderman and Antoni, 2000), can be effectively adapted for our target population of culturally diverse, HIV+, low-income "Recovering Drug Abusers" (RDAs). Since the late 1980s, members of our research team (i.e., Schneiderman, Antoni, Klimas, Fletcher) have been developing, refining and evaluating the effects of CBSM among HIV+ Men who have Sex with Men (MSM). In the early/mid 90s, we began to adapt and evaluate the effects of CBSM in other non-drug abusing subgroups that were emerging with increasing levels of HIV seroprevalence (e.g., pregnant women, African American and Hispanic men and women). After accumulating considerable support for the effectiveness of CBSM in these subgroups in the late 90s, our research team (i.e., Malow, Schneiderman, Antoni, Klimas, Page) turned its attention to developing the CBSM for one of the most neglected and understudied populations affected by the HIV/AIDS epidemic in this country: "inner city" minority drug abusers. With supplemental funding on two NIH grants to conduct formative stage1 pilot research, our project team has been able to develop and document the feasibility and potential promise of the CBSM approach adapted/translated for RDAs (CBSM-RDA). This application proposes to take the next logical step in continuing this work: conducting a 3, 6, 8, 10, and 12 month follow-up outcome study comparing CBSM-RDA with a matched attention, time and interest value Health Promotion Comparison (HPC) condition, in 225 male and 225 female HIV+ RDAs with respect to key biopsychosocial health endpoints: distress (i.e., depressive symptoms, and mood state), quality of life, drug abuse relapse, unsafe sex, Combination Antiretroviral Therapy (CART) medication adherence and health status indicators (e.g., Viral Load, CD4 count, physical symptoms).

DETAILED DESCRIPTION:
The primary purpose of this proposed 5-year study is to determine whether a Cognitive Behavioral Stress Management (CBSM) intervention, demonstrated to be effective in reducing distress, enhancing coping, and maintaining health among HIV+ non-drug abusers (see Schneiderman and Antoni, 2000), can be effectively adapted for our target population of culturally diverse, HIV+, low-income "Recovering Drug Abusers" (RDAs). Since the late 1980s, members of our research team (i.e., Schneiderman, Antoni, Klimas, Fletcher) have been developing, refining and evaluating the effects of CBSM among HIV+ Men who have Sex with Men (MSM). In the early/mid 90s, we began to adapt and evaluate the effects of CBSM in other non-drug abusing subgroups that were emerging with increasing levels of HIV seroprevalence (e.g., pregnant women, African American and Hispanic men and women). After accumulating considerable support for the effectiveness of CBSM in these subgroups in the late 90s, our research team (i.e., Malow, Schneiderman, Antoni, Klimas, Page) turned its attention to developing the CBSM for one of the most neglected and understudied populations affected by the HIV/AIDS epidemic in this country: "inner city" minority drug abusers. With supplemental funding on two NIH grants to conduct formative stage1 pilot research, our project team has been able to develop and document the feasibility and potential promise of the CBSM approach adapted/translated for RDAs (CBSM-RDA). This application proposes to take the next logical step in continuing this work: conducting a 3, 6, 8, 10, and 12 month follow-up outcome study comparing CBSM-RDA with a matched attention, time and interest value Health Promotion Comparison (HPC) condition, in 225 male and 225 female HIV+ RDAs with respect to key biopsychosocial health endpoints: distress (i.e., depressive symptoms, and mood state), quality of life, drug abuse relapse, unsafe sex, Combination Antiretroviral Therapy (CART) medication adherence and health status indicators (e.g., Viral Load, CD4 count, physical symptoms).

ELIGIBILITY:
1. >18, but <60 years of age
2. fluency in spoken English which is required to complete assessments and to participate in the intervention groups;
3. acknowledgement of HIV seropositivity and willingness to be tested to confirm this serostatus;
4. currently not cognitively impaired since cognitive impairment may compromise the ability to comprehend and participate in the assessment and intervention;
5. currently not showing symptoms of a major psychiatric disorder/ including psychosis, or a high risk for suicidality since these conditions might compromise ability to comprehend and participate in the assessment and intervention; and
6. classification as a "Recovering Drug Abusers" (RDAs; 30 days free of substances, 1-36 months recovery from alcohol and other drugs).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450
Dates: Start 1999-09; Study Completion 2007-08

PRIMARY OUTCOMES:
To evaluate if CBSM-RDA produces therapeutic improvement in distress and quality of life indices to a greater extent than HPC.
SPECIFIC AIM 2: To evaluate if CBSM-RDA reduces drug abuse relapse to a greater extent than HPC.
SPECIFIC AIM 3: To evaluate if CBSM-RDA reduces unsafe sex to a greater extent than HPC.
SPECIFIC AIM 4: To evaluate if CBSM-RDA enhances CART adherence to a greater extent than HPC.
SPECIFIC AIM 5: To evaluate if CBSM-RDA enhances health status to a greater extent than HPC.
SPECIFIC AIM 6: To evaluate the extent to which key variables may mediate the relationships between our intervention and endpoints.
SPECIFIC AIM 7: To evaluate the extent to which key variables moderate the relationships between our intervention and endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Malow, PhD, Principal Investigator — Florida International University